CLINICAL TRIAL: NCT07301632
Title: Ecstasy to Alleviate SEvere Chronic Neuropathic Pain (EASE Pain) Trial: A Randomized Controlled Pilot Trial
Brief Title: Ecstasy to Alleviate SEvere Chronic Neuropathic Pain Trial
Acronym: EASEPain
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EASE Pain P-006
Record Dates: First submitted 2025-11-17; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-10

CONDITIONS: Chronic Neuropathic Pain
Keywords: 3, 4-methylenedioxymethamphetamine hydrochloride; Chronic Neuropathic Pain
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine; Methylphenidate

STUDY DESIGN:
Intervention Model Description: Preparatory psychotherapy from week 1 to 5; a single dosing session with psychotherapy at week 6 and integrative psychotherapy at weeks 7 to 16.
  Follow up for primary clinical endpoint and final follow up at week 16.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3,4-Methylenedioxymethamphetamine (Active Comparator): Treatment Arm: 3,4-Methylenedioxymethamphetamine 120mg (3 x 40mg capsule) PO single dose plus psychological support; optional 40mg supplemental dose at 2hr mark if there are no tolerability issues reported, patient consents and lead physician deems appropriate. (Maximum dose 160mg)
  Interventions: Drug: 3,4-Methylenedioxymethamphetamine
- Methylphenidate (Placebo Comparator): Placebo arm: Methylphenidate 30mg (3 x 10mg capsule) PO single dose plus psychological support; optional 10mg supplemental dose at 2hr mark if there are no tolerability issues reported, patient consents and lead physician deems appropriate. (Maximum dose of 40 mg)
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: 3,4-Methylenedioxymethamphetamine — Treatment arm: 3,4-Methylenedioxymethamphetamine 120mg (3 x 40mg capsule) PO single dose plus psychological support; optional 40mg supplemental dose at 2hr mark if there are no tolerability issues reported, patient consents and lead physician deems appropriate. (Maximum dose 160mg)
  Other Names: MDMA
  Arms: 3,4-Methylenedioxymethamphetamine
Drug: Methylphenidate — Placebo arm: Methylphenidate 30mg (3 x 10mg capsule) PO single dose plus psychological support; optional 10mg supplemental dose at 2hr mark if there are no tolerability issues reported, patient consents and lead physician deems appropriate. (Maximum dose of 40 mg)
  Other Names: MDP
  Arms: Methylphenidate

SUMMARY:
This is a Health Canada regulated internal pilot study designed to assess the feasibility, tolerability, and preliminary efficacy of 3, 4-methylenedioxymethamphetamine hydrochloride capsules-AT for chronic neuropathic pain to inform a larger, fully powered multi-center study. This is an interventional, randomized, 2-arm parallel, triple blinded study.

The total study duration is 2 years.

Participants will receive preparatory psychotherapy session during week 2 and week 4 followed by a combined single dosing session with psychotherapy during week 6. Integrative psychotherapy will follow at weeks 6, 8, 12, and 16.

Follow up for primary clinical endpoint at week 16; final follow up for secondary clinical endpoint at 16-weeks.

Participants will be asked to complete adjunctive home psychotherapy in the form of online modules. Data collected will be entered in electronic case report form (REDCap Academic).

DETAILED DESCRIPTION:
Primary objective:

To demonstrate the feasibility of conducting the full EASE Pain trial by achieving targets in recruitment, data completion rate, blinding integrity, minimal serious drug-related adverse events, and by identifying barriers and facilitators to the full trial.

Secondary objectives (full trial):

To evaluate whether a 120 mg dose of oral 3,4-methylenedioxymethamphetamine with an optional 40mg supplementary dose leads to meaningful improvements in pain interference at 16-weeks in patients with moderate-to-severe chronic neuropathic pain compared to active-placebo, and assess changes in physical function, physical activity, emotional function, overall rating of improvement, and adverse events over 16 weeks.

Study type: Intervention trial Allocation: Randomized Intervention model: 2-Arm Parallel Group Primary purpose: Feasibility Phase: Phase II Blinding: Triple blinded (patient- outcome assessor- and psychotherapist-blinded)

Total study duration: 2 years Duration for each subject: 16 weeks. Preparatory psychotherapy from week 1 to 5; a single dosing session with psychotherapy at week 6 and integrative psychotherapy at weeks 7 to 16.

Follow up for primary clinical endpoint and final follow up at week 16.

Dosage regimen:

Treatment arm: 3,4-methylenedioxymethamphetamine 120mg (3 x 40mg capsule) PO single dose plus psychological support; optional 40mg supplemental dose at 2hr mark if there are no tolerability issues reported, patient consents and lead physician deems appropriate. (Maximum dose 160mg)

Placebo arm: Methylphenidate 30mg (3 x 10mg capsule) PO single dose plus psychological support; optional 10mg supplemental dose at 2hr mark if there are no tolerability issues reported, patient consents and lead physician deems appropriate. (Maximum dose of 40 mg)

Treatment/ assessment visits:

Week -1: Screening Week 1: Baseline data collection, psychotherapy workbook 1 (preparation) Week 2: Psychotherapy preparatory session 1 Week 3: Psychotherapy workbook 2 (preparation) Week 4: Psychotherapy preparation session 2 Week 5: Psychotherapy workbook 3 (preparation) Week 6: (Day 0): Randomization to drug and experimental session with in-person psychotherapy (Day 1) Psychotherapy integration session 1 Week7: Psychotherapy workbook 4 (integration). Questionnaire and AE follow up Week 8: Psychotherapy integration session 2 Week 9 to 11 Psychotherapy workbook 5 (integration) Week 10: Questionnaire and AE follow up Week 12: Psychotherapy integration session 3 Week 13 to 15: Psychotherapy workbook 6 (integration) Week 16: Psychotherapy integration session 4. Primary clinical end point (Questionnaires and Adverse Event (AE) follow up)

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults 18 years and older.
* Diagnosis of chronic neuropathic pain (greater than 3 months in duration) by a clinician with specialized training in chronic pain, confirmed with the standardized Leeds Assessment of Neuropathic Symptoms and Signs questionnaire.
* Suffering from moderate-to-severe pain as defined by
* Baseline Patient Reported Outcomes Measurement System - Pain Interference (PROMIS-PI) score of greater than or equal to 60
* An average pain intensity of greater than or equal to 5 on a 0-10 numeric rating scale,43
* Treatment-refractory pain as defined by a failure of ≥2 medications recommended in the Canadian consensus guidelines on the management of CNP to generate self-reported meaningful improvement in symptoms.
* For participants of childbearing potential, use of a highly effective or double-barrier methods of contraception. Abstinence is acceptable if it is the preferred and usual lifestyle of the participant.
* Sufficient English skills to participate in psychotherapy.

Exclusion Criteria:

* Past or current history of a psychotic disorder, mania, hypomania, bipolarity, current suicidal ideation, stimulant use disorder (i.e., cocaine, amphetamine, methamphetamine, MDMA, methylphenidate (Ritalin), etc , and any other substance use disorder within the past 12 months assessed by history and confirmed the Mini-International Neuropsychiatric Interview [MINI]. Other secondary psychiatric comorbidities (e.g., anxiety disorders, trauma related disorders, other personality disorders. etc.) will not be excluded
* Participants with a history of suicide attempts are not excluded unless a significant risk of suicidal behavior is present at the time of screening as determined by the CRSS (Columbia suicide rating scale)
* History of prior MDMA use (excluded to maintain blinding integrity)
* Long QT syndrome, measured by an ECG with a QTc more than 450 ms for males, and 470 ms for females.
* Presence of a relative or absolute contraindication to MDMA or Methylphenidate:
* Pre-existing cardiovascular disorders evidenced in clinical records or disclosed on patient self-report, such as: uncontrolled hypertension (sustained blood pressure ≥160/100 mmHg), angina (ongoing angina at rest, recent hospitalization for acute coronary syndrome within the past 3 months, or a history of revascularization (e.g., stenting or bypass surgery) within the past 6 months), arterial occlusive disease; heart failure, hemodynamically significant congenital heart disease, cardiomyopathies, myocardial infarction (within the past 6 months), potentially life-threatening arrhythmias (new-onset within the last 3 months), arrhythmias causing hemodynamic instability (SBP < 90 mm Hg), or requiring urgent intervention (e.g., atrial fibrillation with rapid ventricular response or ventricular tachycardia), channelopathies, aneurysmal vascular disease (e.g., thoracic and/or abdominal aorta, intracranial, and peripheral arterial vessels), advanced arteriosclerosis
* Cerebrovascular conditions: acute stroke or recent history of intracerebral hemorrhage (ischemic or hemorrhagic stroke occurring within the past 6 months)
* Conditions at risk of elevation of blood pressure and increase heart rate, such as glaucoma, tension, agitation, thyrotoxicosis, pheochromocytoma
* Motor tics and/or family history or diagnosis of Tourette's syndrome
* Moderate to severe chronic kidney disease or kidney failure, such as requiring dialysis, significant treatment adjustments for kidney function, or regular nephrologist follow-up)
* Moderate to severe liver disease, such as cirrhosis, a history of significant jaundice unrelated to temporary illness, or any liver condition requiring regular monitoring by a specialist).
* Current treatment with selective serotonin reuptake inhibitors (SSRI's) and serotonin-norepinephrine reuptake inhibitors (SNRI's), tricyclic antidepressants, serotonin 5-HT1 receptor agonists (triptans) and 5-HT3 receptor antagonist antiemetics (risk of Serotonin Syndrome)
* Hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption (methylphenidate contains lactose)
* Seizure disorders
* Pregnancy, or breastfeeding
* Known hypersensitivity to study drugs or any study drug excipients
* Medications that interact with study drugs including:
* Any lifetime history use of any stimulant medication (e.g., Adderall, Vyvanse, Ritalin)
* Caffeine intake within 24 hours
* Monoamine oxidase inhibitors (MAOI) within 14 days (e.g. phenelzine, moclobemide, isoniazid, linezolid, phenelzine, harmine) due to risk of hypertensive crisis
* CYP2D6 substrates and modifiers (such as: buproprion, fluoxetine, paroxetine, duloxetine, mirabegron).
* Adrenergic agents (e.g. clonidine) risk of sudden death
* Vasopressor agents (ephedrine pseudoephedrine)
* Coumarin anticoagulants (e.g., warfarin),
* Anticonvulsants (e.g., phenobarbital, diphenylhydantoin, primidone)
* Anti-psychotics and inhibitors of dopamine uptake (e.g. haloperidol, DOPA, tricyclic antidepressants)
* Concomitant medication that could prolong ECG QT interval (e.g. ondansetron, risperidone, methadone)
* Selective Serotonin Reuptake Inhibitors (citalopram, sertraline, fluvoxamine, escitalopram)
* Selective Norepinephrine Uptake Inhibitors (e.g. venlafaxine, duloxetine); Serotonergic Drugs (e.g. dextromethorphan, fentanyl, St. John's Wort, tramadol, 5-hydroxytryptophan); serotonin 5-HT1 receptor agonists (triptans) and 5-HT3 receptor antagonist antiemetics due risk of Serotonin Syndrome which is a potentially life- threatening condition
* Currently engaged in psychotherapy for CNP (other psychotherapy for non-CNP is allowed).
* Any other clinically significant medical illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if they take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-17 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this pilot trial is to determine feasibility of a large-scale, multi-center trial. | 16 weeks
  Average Monthly recruitment of >1 participant per center means that the full trial should meet recruitment requirements within 12 months.
Secondary feasibility outcome | 16 weeks
  Data completion rate (of primary clinical outcome)≥ 80%
Participant Retention | 16 weeks
  Retention of ≥80% of participants at the reported primary outcome point of 16 weeks after the experimental session should minimize attrition bias in the definitive trial's primary outcome data (e.g. withdrawal due to side-effects)
Blinding | 16 weeks
  Blinding Integrity (≤80% of participants in both arms correctly guess their treatment allocation (Note: 50% of participants would be expected to correctly guess treatment allocation due to chance alone)
Adverse Events | 16 weeks
  ≤3 serious drug-related adverse events
Secondary Feasibility Outcome | 16 weeks
  identification of patient, clinician and researcher-identified trial barriers using qualitative methods (e.g. interviews at the end of the study with participants who provides consent )

SECONDARY OUTCOMES:
The Patient-Reported Outcomes Measurement Information System (PROMIS) pain Intensity, Pain Interference and Physical Function Scale | Week 1, Week 7, Week 11 and Week 16
  In the past 7 days patients to rate their pain on average- 0 scale-indicates No pain and 10 scale- indicates Worst imaginable pain
Patient Health Questionnaire (PHQ-9) | Week 1, Week 7, Week 11 and Week 16
  Over the last 2 weeks how often the patient has been bothered by daily activities on a scale of 0 to 3. 0 (Not at all) and 3 (Nearly every day)
Generalized Anxiety Disorder 7-Item (GAD-7) Questionnaire | Week 1, Week 7, Week 11 and Week 16
  Over the last 2 weeks, how often patients have been bothered by anxiety on a scale of 0 to 3. 0 equals Not at all and 3 equals Nearly every day
The Post traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual for Mental Disorder-5 (PCL-5) | Week 1, Week 7, Week 11 and Week 16
  Over the past month, how patients were bothered by internal and external feelings like stress, negativity etc. This is measured on a scale of 0 (Not at all) to 4 (Extremely)
Health Questionnaire (EQ-5D-5L) | Week 1, Week 7, Week 11 and Week 16
  Patients to describe how their health is affected in terms of mobility, self-care, Usual activities like (work, study, family), Pain/Discomfort, Anxiety/Depression on a scale of 0( Worst health you can imagine) to 100 (Best health you can imagine)
The Patient Global Impression of Change Scale (PGIC) | Week 7, Week 11 and Week 16
  This questionnaire measures how the patient impression changed before being enrolled in the study. Measured in a scale of 1 (Very much Improved) to 7 ( Very Much Worse)
The Toronto Side Effect Scale (TSES) | Week 7, Week 11 and Week 16
  This questionnaire measures patient's symptoms in the last two weeks for Agitation, tremor, twitching etc in terms of frequency and Severity in a scale of 1 (Never) to 5 (Every day)
STAR-P | Week 7, Week 11 and Week 16
  This questionnaire measures patient's perception and attitude regarding the clinician on a scale of 0 (Never) to 4 (Always)
Subjective Drug Effects (VAS) | Week 6
  On a scale of 0 (Not at all) to 10 (Extremely) patients to describe their experience during intervention session regarding the subjective drug effects

CONTACTS AND LOCATIONS:
Overall Officials: Akash Goel, MD,MPH,FRCPC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada